CLINICAL TRIAL: NCT02521337
Title: PreTerm RNA in Maternal Serum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Pre Term MiRNA-HMO-CTIL
Record Dates: First submitted 2015-07-12; First posted 2015-08-13 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- pregnant women not in active labor
  Interventions: Other: observation
- pregnant women in preterm labor
  Interventions: Other: observation
- pregnant women in term labor
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
Preterm birth is defined as a birth occurring before the completion of 37 weeks gestation. The incidence of preterm birth in Israel in the last years is around 7-8%.

Despite various diagnostic modalities as well as newly therapeutic approaches the incidence of preterm birth remains unchanged and is considered to be the leading cause of neonatal morbidity and mortality.

In the last decade, small RNAs have emerged as an important player in both physiological and pathophysiological responses. These single strands, non-coding regulatory RNA molecules are responsible for post transcriptional regulation of target genes. Hence, may provide a new opportunity for biomarkers discovery in the field of preterm birth.

The main objective of this study is to identify a distinctive expression profile of maternal circulating RNAs that will be used as biomarkers for preterm birth.

ELIGIBILITY:
Inclusion Criteria:

1. Women with singleton pregnancy at 26-32 week of gestation with no clinical symptoms of preterm labor.
2. Women with singleton pregnancy 24-34 week of gestation who present to the labor suite with symptoms suspected for preterm labor.
3. Women with singleton pregnancy in term active labor (weeks 37-40).

Exclusion Criteria:

Exclusion criteria will include:

1. multiple gestation,
2. major fetal anomalies,
3. IUFD,
4. severe preeclampsia,
5. chronic steroid or immunosuppressive drug use,
6. active immunological illness,
7. and/or pregestational and gestational DM.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of women with preterm labor that present a unique RNA cluster | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel